CLINICAL TRIAL: NCT04551924
Title: A Phase I Study to Evaluate the Safety, Pharmacokinetics and Efficacy of HR18034 for Pain Management After Inguinal Hernia Repair
Brief Title: A Trial of HR18034 in Inguinal Hernia Repair
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HR18034-101
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Inguinal Hernia Repair
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain objectiveness, the study drug will be managed and administered by an independent unblinded team. Subjects, investigators, and all other site staff who directly interact with subjects, evaluate safety and efficacy, and collect subject data, will remain blinded and must not communicate or discuss any study information with the unblinded team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- dose 1 (Experimental): HR18034（Ropivacaine Liposome for Injection） is a sustained-release liposome
  Interventions: Drug: HR18034
- dose 2 (Experimental): HR18034（Ropivacaine Liposome for Injection） is a sustained-release liposome
  Interventions: Drug: HR18034
- dose 3 (Experimental): HR18034（Ropivacaine Liposome for Injection） is a sustained-release liposome
  Interventions: Drug: HR18034
- dose 4 (Experimental): HR18034（Ropivacaine Liposome for Injection） is a sustained-release liposome
  Interventions: Drug: HR18034
- Naropin (Active Comparator): Naronpin injection contains ropivacaine HCl. Strength: 150mg/ 30mL (5 mg/mL) Size: 30mL fill, in a 30mL single dose vial
  Interventions: Drug: Naropin

INTERVENTIONS:
Drug: HR18034 — HR18034（Ropivacaine Liposome for Injection） is a sustained-release liposome
  Other Names: subjects will receive HR18034.
  Arms: dose 1; dose 2; dose 3; dose 4
Drug: Naropin — Local infiltration of Naropin to produce anesthesia for surgery and analgesia in postoperative pain management. Naropin 150mg [0.5%, 5mg/mL] x 30mL
  Other Names: Naropin, 0.5% Injectable Solution
  Arms: Naropin

SUMMARY:
Phase I, randomized, double-blind, comparator-controlled study to assess the safety, PK, and efficacy of single postsurgical application of HR18034 compared with Naropin®

ELIGIBILITY:
Inclusion Criteria:

Able and willing to provide a written informed consent 2、Male or female between 18 and 70 years of age 3、Scheduled to undergo a primary, inguinal hernia repair with mesh, and be able to use the anesthesia regimen 4、Meet the body mass 5、Conform to the ASA Physical Status Classification

Exclusion Criteria:

1. Clinically significant abnormal clinical laboratory test value
2. Subjects with poor blood pressure control after medication
3. Subjects with atrioventricular block or cardiac insufficiency
4. Subjects with a history of myocardial infarction or unstable angina pectoris
5. Subjects with a history of ischemic stroke or transient ischemic attack
6. Combination of other pain conditions that may affect postoperative pain assessment
7. Allergic to a drug ingredient or component
8. Persistent or recurrent nausea and/or vomiting due to other etiologies, including, but not limited to gastric outlet obstruction, hypercalcemia, or active peptic ulcer
9. History of alcohol abuse or prescription and/or illicit drug abuse within 1 years
10. Subjects with special diets (including tobacco, grapefruit and caffeine)
11. Positive results on the urine drug screen or alcohol breath test indicative of illicit drug or alcohol abuse.
12. History of human immunodeficiency virus (HIV), hepatitis C, syphilis antibody，or hepatitis B.
13. Use of any of the following medications within 14 days or as specified prior to the study surgical procedure:
14. Have had an inguinal hernia repair in the last 3 months before the study surgical procedure or presents with bilateral or recurrent inguinal hernia, other hernia presentations, or hernias with a large scrotal component that would be difficult to reduce surgically
15. Participated in clinical trials of other drugs (received experimental drugs)
16. History or clinical manifestations of significant renal, hepatic, gastrointestinal, cardiovascular, metabolic, neurologic, psychiatric, or other condition.
17. Pregnant or nursing women
18. No birth control during the specified period of time
19. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of SAEs and treatment-related severe AEs | 14 days
  Safety and tolerability:

SECONDARY OUTCOMES:
Pain intensity assessed using an 11-point NPRS ranging | Baseline till 168 hours post IP administration
  11-point Numercal Pain Rating Scale ranging from a score of 0 to 10. Pain-free defined as an NPRS of 0 or 1. Worst imaginable pain defined as an NPRS of 10
AUC of NPRS | For time periods 0-12, 0-24, 0-36, 0-48, 0-72, and 0-96 hours
  AUC of NPRS for time periods 0-12, 0-24, 0-36, 0-48, 0-72, and 0-96 hours
Patient Global Assessment of the method of pain control | 24 hours post IP administration till 168 hours post IP administration
  Patient Global Assessment ranging from a score of 0 to 10. Satisfaction defined as a scale of 10, dissatisfaction defined as a scale of 0.
Proportion of pain-free subjects at scheduled timepoints. | Baseline till 168 hours post IP administration
  Pain-free defined as an NPRS of 0 or 1
Proportion of subjects who used no rescue opioid analgesic | Baseline till 168 hours post IP administration
  Proportion of subjects who used no rescue opioid analgesic
Average daily rescue analgesic consumption | Baseline till 168 hours post IP administration
  Average daily rescue analgesic consumption through 24, 48, 72 and 96 hours
Time to the first postoperative use of rescue opioid analgesics | Baseline till 168 hours post IP administration
  Time to the first postoperative use of rescue opioid analgesics
PK Cmax | Baseline till 168 hours post IP administration
  Maximum blood concentration (Cmax)
Wound assessment by Wound healing and status score | Day 1 through Day 14
  The surgical site will be examined by the investigator using Wound healing and status score. Wound healing and status score ranging from a score of 0 to 4，Good defined as a scale of 0. Worst defined as a scale of 4.
PK AUC | Baseline till 168 hours post IP administration
  Area under the blood concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China